CLINICAL TRIAL: NCT01908478
Title: A Phase I Study of Veliparib (ABT-888) in Combination With Gemcitabine and Intensity Modulated Radiation Therapy in Patients With Locally Advanced, Unresectable Pancreatic Cancer
Brief Title: Veliparib in Combination With Gemcitabine and Intensity Modulated Radiation Therapy in Patients With Pancreatic Cancer
Acronym: VelGemRad
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Richard Tuli, MD, Assistant Professor, Radiation Oncology, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS-ABT888-0002
Record Dates: First submitted 2013-07-18; First posted 2013-07-25 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Cancer
Keywords: locally advanced; unresectable; pancreatic; pancreas; pancreatic adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — veliparib; Gemcitabine; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination: veliparib, gemcitabine, and IMRT (Experimental)
  Interventions: Drug: Veliparib; Drug: Gemcitabine; Radiation: Intensity modulated radiation therapy

INTERVENTIONS:
Drug: Veliparib
  Other Names: ABT-888
Drug: Gemcitabine
  Other Names: Gemzar
Radiation: Intensity modulated radiation therapy

SUMMARY:
This is a Phase I Study of veliparib (ABT-888) in combination with Gemcitabine and Intensity Modulated Radiation Therapy in Patients with Locally Advanced, Unresectable Pancreatic Cancer.

Primary Objectives:

* Determine the maximum tolerable dose of veliparib in combination with gemcitabine and intensity modulated radiation therapy in patients with locally advanced pancreatic cancer.
* Determine the safety and toxicity of the combination of veliparib with gemcitabine and radiation therapy in patients with locally advanced pancreatic cancer

DETAILED DESCRIPTION:
Gemcitabine will be administered by intravenous infusion of 1000 mg/m2 over 30 minutes on days 1, 8, 15 of the cycle. Intensity modulated radiation therapy (IMRT) will be given to a total dose of 36 Gy in 15 fractions (2.4 Gy per fraction, one fraction per day, 5 fractions per week, Monday through Friday) beginning on day 1. Veliparib will be administered per a dose escalation schema. The starting dose of veliparib is 20 mg BID based upon safety/efficacy data available. Dose escalation will continue in 20 mg increments until the maximum tolerated dose (MTD) is reached. Intra-patient dose escalation will not be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathological or cytological diagnosis of adenocarcinoma of the pancreas, as well as those with high clinical suspicion of adenocarcinoma, which is deemed locally advanced unresectable or borderline resectable as determined by a pancreatic cancer surgeon and/or following evaluation by a GI oncology tumor board.
* Age 18 years or older

Exclusion Criteria:

* Patients who have had prior anti-cancer treatment for their disease
* Patients who are currently receiving any other investigational agents
* Metastatic disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PARP [Poly (ADP-ribosome) polymerase] inhibitors or gemcitabine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of veliparib based on the incidence of dose-limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I) | Days 1-70

SECONDARY OUTCOMES:
Assessment of objective response rates measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | From baseline to Week 26
  Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response
Evaluation of pre-treatment biopsy specimens for levels of various DNA repair proteins | Baseline only
Change in PAR [Poly(ADP-ribosyl)ation] levels in peripheral blood mononuclear cells | Baseline, Weekly for 6 weeks, and at Weeks 10, 18, and 26

CONTACTS AND LOCATIONS:
Overall Officials: Richard Tuli, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States